CLINICAL TRIAL: NCT02168400
Title: Combining Neuro-Imaging and Non-Invasive Brain Stimulation for Clinical Intervention in Alcohol Use Disorder
Brief Title: Clinical Intervention in Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSYCH-2016-22561; K01AA026349 (NIH)
Record Dates: First submitted 2014-06-13; First posted 2014-06-20 (Estimated); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use Disorder; Eligible to go Into the MRI Scanner; Short-term Abstinence From Alcohol Use (2 Week Abstinent)
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active tDCS (Experimental): Subjects that are randomly assigned to this arm will receive 10 active transcranial direct current stimulation (tDCS) sessions
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- sham tDCS (Sham Comparator): Subjects randomly assigned to sham-tDCS (transcranial direct current stimulation) will receive very low current stimulation at beginning and end of session, mimicking the feeling of current stimulation in the scalp, but not reaching levels that will stimulate brain function.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS will be performed with Neuroelectrics Starstim Enobio 20, a non-invasive investigational device that has been labeled as a non-significant risk device by the FDA. This study is regulated by the FDA as an Abbreviated IDE. It has built-in safety mechanisms which allow for immediate cessation of stimulation if the subject becomes uncomfortable. The current will be administered via two electrode sponges for 25 mins with 1-2 milliamperes. These administration protocols are in line with protocols that have outlined safe administration (Nitsche 2007; 2008). No side-effects have been reported with the exception of slight itching under the electrode and occasional occurrence of headache, fatigue, or nausea (Poreisz 2007). Electrodes placement: dorsolateral prefrontal cortex (DLPFC); cathode on left DLPFC, anode on right DLPFC.
  Other Names: Starstim

SUMMARY:
Long-term abstinence from alcohol is supported by a compensatory mechanism in functional brain connectivity, a potential brain biomarker that could be an intervention target. These findings provide a compelling case to explore whether this brain biomarker can be modulated to enhance patients' ability to remain abstinent. There is a need to investigate methods that can be used to increase functional brain connectivity. The overall objective of this proposal is to enhance brain functional connectivity in short-term abstinent alcoholics as a therapeutic intervention that supports abstinence.

DETAILED DESCRIPTION:
The relapsing nature of alcoholism is a major obstacle to successful treatment. About 60% of those entering treatment will relapse within one year. To improve treatment outcome, new interventions targeting the underlying brain biomarkers of relapse vulnerability hold significant promise in reducing this critical public health problem. Using resting functional magnetic resonance imaging (fMRI) the investigators have identified brain biomarkers that support long-term abstinence. Cross-sectional and longitudinal findings provide evidence that higher functional connectivity (FC), particularly between nucleus accumbens (NAcc) and dorsolateral prefrontal cortex (DLPFC), is a potential brain biomarker that supports abstinence. Long-term abstinent alcoholics (7 years of abstinence) have higher resting FC between NAcc and DLPFC when compared to controls. Short-term abstinent alcoholics (11 weeks of abstinence) have intermediate FC (lower than long-term abstinent alcoholics and higher than controls). Further, lower FC between NAcc and DLPFC at 11 weeks of abstinence can be a predictor of subsequent relapse (with 74% accuracy). Moreover, in a pilot longitudinal FC study examining resting FC of NAcc at 5 and 13 weeks of abstinence in individuals with substance use disorder, the investigators found that FC between NAcc and DLPFC decreased from 5 to 13 weeks of abstinence in subsequent relapsers, while it increased in subsequent abstainers. Based on the above, the investigators believe that long-term abstinence is supported by a compensatory mechanism that mediates proper executive function over reward (mediated by PFC-NAcc FC), a potential brain biomarker that could be an intervention target. These findings provide a compelling case to explore whether this brain biomarker can be modulated to enhance patients' ability to remain abstinent. There is a need to investigate methods that can be used to increase FC between DLPFC and NAcc.

Cognitive flexibility, the ability to change maladaptive behavior, depends on DLPFC input to NAcc. DLPFC transmits reward representations to NAcc through glutamatergic projections that guide goal-directed behavior. If DLPFC fails to activate when required, a common observation in substance use disorder, target neurons in the NAcc core do not receive critical information needed to select the appropriate outcome, causing acquired maladaptive response patterns to persist (e.g. drug consumption). Higher FC between DLPFC and NAcc may be achieved by stimulating DLPFC while subjects perform a task that requires cognitive flexibility, the reversal learning task.

Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that can modulate brain connectivity. DLPFC stimulation may increase input to NAcc to facilitate proper selection of goal-directed behavior and may also decrease craving in individuals with substance use disorder.

Genetics and treatment response: A source of treatment response variability could stem from differences between participants in baseline genetic profiles or epigenetic changes over the course of treatment. Genetic polymorphisms, especially in genes important for neuroplasticity, may also mediate neuroplastic changes underlying the effects of tDCS, as has been demonstrated with gene BDNF. In light of these genetic influences on key tenants of the study - i.e. treatment response in alcohol use disorder and psychological effects of tDCS - the investigators will collect genetic samples from participants to determine whether genetic or epigenetic variations may affect response to the cognitive training and tDCS intervention. As the secondary aim, participants will be given the choice in the consent form to opt in or out of the genetic sampling procedure.

In a double-blind randomized design, up to 100 abstinent (2 weeks abstinent) individuals with alcohol use disorder (AUD) recruited from Lodging Plus Program will receive 10 sessions (2 sessions per day for 5 days) of either (i) transcranial direct current stimulation (tDCS) to PFC or (ii) sham-tDCS. All subjects will perform the reversal learning task during tDCS intervention (active or sham) to prime the engagement of the NAcc-PFC brain circuit that mediates cognitive flexibility. Rest fMRI and craving measures will be collected before the first and after the last day of tDCS sessions. Monthly follow-up interviews will be conducted for 6 months after study completion to query relapse status. Dependent variables will be (i) change in NAcc-PFC FC between 2 and 3 weeks of abstinence, (ii) change in craving scores between 2 and 3 weeks of abstinence and (iii) relapse status ~8 months after study participation. Aim 1: To investigate whether NAcc-PFC FC can be modulated, the investigators will compare magnitude and durability of change in NAcc-PFC FC between active-tDCS and sham-tDCS groups. Aim 2: To determine if PFC stimulation has a short-term effect on behavior related to clinical outcome, the investigators will compare change in craving scores (difference in craving scores between 2 and 3 weeks of abstinence) between active-tDCS and sham-tDCS groups. Aim 3: To correlate neuromodulation intervention with long-term clinical outcome, the investigators will record craving and relapse status during the ~8 months following treatment discharge. The investigators will examine the relationship between change in NAcc-PFC FC between 2 and 3 weeks of abstinence and subsequent (i) monthly craving scores and (ii) relapse status. Aim 4: Examine relationship between genetic variants, epigenetic changes and treatment outcome (e.g. durability, functional connectivity).

ELIGIBILITY:
Inclusion Criteria:

* up to 75 abstinent individuals (18-65 years old; 2 weeks of abstinence) who meet DSM-V criteria for alcohol use disorder (AUD) will be recruited from the Lodging Plus Program, part of University of Minnesota Medical Center
* This 28-day program provides a supervised environment to treat alcoholism in which patients receive random drug/alcohol screenings daily. Lodging Plus has 50 beds and admits an average of 20 patients per week and 59% of patients admitted have a diagnosis of alcohol use disorder.

Inclusion criteria:

* ability to provide written consent and comply with study procedures
* meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnostic criteria for AUD. Subjects may have current comorbid drug use, but their primary substance use disorder diagnosis needs to be based on alcohol use. Subjects must have the intention to remain in program until the end of the study (3 weeks). Vulnerable populations will not be included

Exclusion Criteria:

* any medical condition or treatment with neurological sequelae (i.e. stroke, tumor, loss of consciousness of more than 30 min, HIV)
* a head injury resulting in a skull fracture or loss of consciousness exceeding 30 minutes (i.e., moderate or severe TBI)
* any contraindications for tDCS or MRI scanning (tDCS contraindications: history of seizures; MRI contraindications; metal implants, pacemakers or any other implanted electrical device, injury with metal, braces, dental implants, non-removable body piercings, pregnancy, breathing or moving disorder.)
* any primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder). Participants with other treated and stable psychiatric disorders will be included.
* presence of a condition that would render study measures difficult or impossible to administer or interpret
* age outside the range of 18 to 65
* primary current substance use disorder diagnosis on a substance other than alcohol except for caffeine or nicotine
* clinical evidence of Wernicke-Karsakoff syndrome
* left handedness
* entrance to the treatment program. under court mandate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jazmin Camchong, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Camchong J, Macdonald AW 3rd, Mueller BA, Nelson B, Specker S, Slaymaker V, Lim KO. Changes in resting functional connectivity during abstinence in stimulant use disorder: a preliminary comparison of relapsers and abstainers. Drug Alcohol Depend. 2014 Jun 1;139:145-51. doi: 10.1016/j.drugalcdep.2014.03.024. Epub 2014 Mar 29. PMID 24745476
- [Background] Camchong J, Stenger A, Fein G. Resting-state synchrony during early alcohol abstinence can predict subsequent relapse. Cereb Cortex. 2013 Sep;23(9):2086-99. doi: 10.1093/cercor/bhs190. Epub 2012 Jul 20. PMID 22819968
- [Background] Camchong J, Stenger VA, Fein G. Resting-state synchrony in short-term versus long-term abstinent alcoholics. Alcohol Clin Exp Res. 2013 May;37(5):794-803. doi: 10.1111/acer.12037. Epub 2013 Feb 19. PMID 23421812
- [Background] Ballard K, Knutson B. Dissociable neural representations of future reward magnitude and delay during temporal discounting. Neuroimage. 2009 Mar 1;45(1):143-50. doi: 10.1016/j.neuroimage.2008.11.004. Epub 2008 Nov 24. PMID 19071223
- [Background] Boggio PS, Sultani N, Fecteau S, Merabet L, Mecca T, Pascual-Leone A, Basaglia A, Fregni F. Prefrontal cortex modulation using transcranial DC stimulation reduces alcohol craving: a double-blind, sham-controlled study. Drug Alcohol Depend. 2008 Jan 1;92(1-3):55-60. doi: 10.1016/j.drugalcdep.2007.06.011. Epub 2007 Jul 19. PMID 17640830
- [Background] D'Cruz AM, Ragozzino ME, Mosconi MW, Pavuluri MN, Sweeney JA. Human reversal learning under conditions of certain versus uncertain outcomes. Neuroimage. 2011 May 1;56(1):315-22. doi: 10.1016/j.neuroimage.2011.01.068. Epub 2011 Jan 28. PMID 21281720
- [Background] Gruber AJ, Hussain RJ, O'Donnell P. The nucleus accumbens: a switchboard for goal-directed behaviors. PLoS One. 2009;4(4):e5062. doi: 10.1371/journal.pone.0005062. Epub 2009 Apr 7. PMID 19352511
- [Background] Klauss J, Penido Pinheiro LC, Silva Merlo BL, de Almeida Correia Santos G, Fregni F, Nitsche MA, Miyuki Nakamura-Palacios E. A randomized controlled trial of targeted prefrontal cortex modulation with tDCS in patients with alcohol dependence. Int J Neuropsychopharmacol. 2014 Nov;17(11):1793-803. doi: 10.1017/S1461145714000984. Epub 2014 Jul 10. PMID 25008145
- [Background] Lang N, Siebner HR, Ward NS, Lee L, Nitsche MA, Paulus W, Rothwell JC, Lemon RN, Frackowiak RS. How does transcranial DC stimulation of the primary motor cortex alter regional neuronal activity in the human brain? Eur J Neurosci. 2005 Jul;22(2):495-504. doi: 10.1111/j.1460-9568.2005.04233.x. PMID 16045502
- [Background] Monte-Silva K, Kuo MF, Hessenthaler S, Fresnoza S, Liebetanz D, Paulus W, Nitsche MA. Induction of late LTP-like plasticity in the human motor cortex by repeated non-invasive brain stimulation. Brain Stimul. 2013 May;6(3):424-32. doi: 10.1016/j.brs.2012.04.011. Epub 2012 Jun 2. PMID 22695026
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Nitsche MA, Doemkes S, Karakose T, Antal A, Liebetanz D, Lang N, Tergau F, Paulus W. Shaping the effects of transcranial direct current stimulation of the human motor cortex. J Neurophysiol. 2007 Apr;97(4):3109-17. doi: 10.1152/jn.01312.2006. Epub 2007 Jan 24. PMID 17251360
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 consented participants were not randomized to either study group and were excluded from the study
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 39 | 36
Completed | 31 | 29
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 39 | 36 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 36 | 75
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.66 (10.43) | 43.31 (9.95) | 41.87 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 27 | 24 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 31 | 25 | 56
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Intervention Effects on Brain Functional Connectivity
Description: Compared mean change in brain functional connectivity (measured at two timepoints, at pre-intervention and at post-intervention) between Active tDCS and Sham groups.
Time Frame: 1 week
Measure: Mean (Standard Error); unit: percentage of Blood Oxygenation Level De
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 31 | 29
percentage of Blood Oxygenation Level De | 0.05 (0.05) | 0.19 (0.19)

2. Secondary Outcome: Correlation Between Functional Connectivity Change and Clinical Outcome (Length of Abstinence)
Description: Pearson correlation, X variable was change in functional connectivity as defined by connectivity from dorsolateral prefrontal cortex to incentive salience network, Y variable was clinical outcome as defined by length of abstinence after intervention.
Time Frame: 8 months
Measure: Mean (Standard Error); unit: correlation coefficient
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 31 | 29
correlation coefficient | 0.03 (0.07) | 0.16 (0.2)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/39 | 1/36
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/36
Other Adverse Events (participants affected / at risk) | 0/39 | 2/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS (N=39) | Sham tDCS (N=36)
Hair loss (not associated with study, MD identified hair loss was due to malnutrition) (General disorders) | 0 (0) | 1 (1)
Mood changes (not associated with research study, participant had prexisting mood disorder) (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT02168400/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT02168400/ICF_001.pdf